CLINICAL TRIAL: NCT01294618
Title: "Phase II Multicenter Study Evaluating the Efficacy and the Safety of a Combination of Nilotinib Plus Pegylated Interferon Alpha 2a for de Novo Chronic Phase Chronic Myelogenous Leukemia Patients"
Brief Title: Nilotinib + Pegylated Interferon Alpha 2a for Untreated Chronic Phase Chronic Myelogenous Leukemia
Acronym: NILOPEG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-560
Record Dates: First submitted 2011-02-07; First posted 2011-02-11 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2011-02

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Chronic Myelogenous Leukemia; nilotinib; pegylated interferon; BCR-ABL Philadelphia chromosome; Hematologic, cytogenetic and molecular response rates and kinetics will be studied in addition to the safety of the combination
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nilotinib + pegylated interferon alpha 2a (PEG-IFN). (Experimental)
  Interventions: Drug: Nilotinib,Novartis,300 mg twice a day +Pegylated interferon 2a,Roche, 45 microg weekly starting Month 2-Month 12 or beyond according to investigator choice.

INTERVENTIONS:
Drug: Nilotinib,Novartis,300 mg twice a day +Pegylated interferon 2a,Roche, 45 microg weekly starting Month 2-Month 12 or beyond according to investigator choice. — Combination of both treatments active by different means on the leukemic cells, in order to enhance the response rates of CP CML patients since diagnosis.

SUMMARY:
The aim of this study is to demonstrate the safety and the efficacy of a combination of 2 treatments shown to have some efficacy in Chronic Phase Chronic Myelogenous Leukemia (CP CML) separately, but that have never been combined to date, and this combination is expected to substantially increase the molecular response rates.

ELIGIBILITY:
Inclusion Criteria:

* Performans status 0-2
* CP CML diagnosed since less than 3 months without previous Tyrosine Kinase Inhibitor (TKI) or interferon treatment
* Adequate organic functions:

  * Total Bilirubin < 1.5xUpper Normal Range (UNR).
  * Aspartate Amino Transferase (ASAT) and Alanine Amino Transferase (ALAT) < 2.5xUNR.
  * Alkaline phosphatase ≤ 2.5xUNR
  * Amylase and lipase ≤ 1.5xUNR.
  * Creatininemia < 1.5xUNR.
* Biological blood standards :

  * Potassium ≥ Lower Normal Range (LNR)
  * Magnesium ≥ LNR.
  * Phosphorus ≥ LNR
  * Calcium ≥ LNR.
* Negative pregnancy test within the last 7 days for women with childbearing potential.
* Informed consent signed up
* Compliance to tretament ensured,
* Valid social insurance

Exclusion Criteria:

Prior TKI or interferon treatment for the CML

* Contra-indication to IFN
* Pregnancy, breast feeding
* Human Immunodeficiency Virus positive, chronic hepatitis B or C.
* Other BCR-ABL transcript than M-bcr
* Cardiopathy defined as:

  * Left Ventricular Ejection Fraction (LVEF) < 45%.
  * Left bundle branch block
  * Ventricular pacemaker.
  * Congenital prolonged QT
  * Past ventricular or significant auricular tachyarrythmia
  * Clinically significant bradycardia (<50 per minute).
  * QTc (Fredericia) > 450 ms (average on 3 Elektrokardiogramm (EKG)).
  * Myocardial infarction in the last 12 months.
  * Unstable angina within the last 12 months.
  * Other significant cardiac diseases.
* Other uncontrolled severe disease (such as diabetes melittus etc…)
* Other ongoing malignant disease.
* Past history of congenital or acquired clinically significant bleeding disorder.
* Previous radiotherapy ≥25% of bone marrow.
* Serious surgery within the past 4 weeks
* Investigational treatment within the last 30 days prior to day 1.
* History of non compliance.
* Cytochrome P450 3A4 (CYP3A4) inhibitors that could not be withdrawn or modified (such as erythromycin, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, ritonavir, mibefradil).
* Severe gastro-intestinal disorders (such as gastric ulcer, uncontrolled nausea, malabsorption syndrome, small intestine resection, gastric shunt).
* Hepatic, renal or pancreatic chronic disorder unrelated to CML
* Recent history of acute pancreatitis within a year or history of chronic pancreatic disease .
* Any concommittant treatment inducing QT prolongation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of complete molecular remissions after 12 months of treatment with nilotinib + Pegylated Interferon (PEG-IFN) | 24 months
  The trial opens for enrolment in 2011 March 7th for 18 months. Each patient will be followed for 24 months after entry.

SECONDARY OUTCOMES:
Kinetics of Complete Molecular Response (CMR) at 1, 2, 3, 6, 9, 12, 15, 18 and 24 months. | Patients will be enrolled for 18 months and will be followed for 24 months
  CMR corresponds to a level of BCR-ABL transcripts < 0.001 % (BCR-ABL/ABL ratio < 0.001%). The BCR-ABL/ABL ratio will be analysed by Reverse Transcription Polymerase Chain Reaction (RT-PCR) at 1, 2, 3, 6, 9, 12, 15, 18 and 24 months to study kinetics of CMR.
Stability of CMR : Proportion of patients maintaining their CMR at 18 and 24 months | Patients will be enrolled for 18 months and will be followed for 24 months
Kinetics of Major Molecular Response (MMR) at 1, 2, 3, 6, 9, 12, 15, 18 and 24 months. | Patients will be enrolled for 18 months and will be followed for 24 months
  MMR corresponds to a level of BCR-ABL transcripts < 0.1 % (BCR-ABL/ABL ratio < 0.1%). The BCR-ABL/ABL ratio is analysed by RT-PCR at 1, 2, 3, 6, 9, 12, 15, 18 and 24 months to study kinetics of MMR.
Stability of MMR : proportion of patients maintaining their MMR at 18 and 24 months | Patients will be enrolled for 18 months and will be followed for 24 months
Cumulative Complete Cytogenetic Remission (CCyR) rates at 3, 6 and 12 months. | Patients will be enrolled for 18 months and will be followed for 24 months
Safety (hematologic and non-hematologic) of the combination nilotinib + PEG-IFN | Patients will be enrolled for 18 months and will be followed for 24 months
Dose reductions or interruptions of each treatment studied | Patients will be enrolled for 18 months and will be followed for 24 months
Progression free survival. | Patients will be enrolled for 18 months and will be followed for 24 months
Overall survival. | Patients will be enrolled for 18 months and will be followed for 24 months
Quality of life on nilotinib + PEG-IFN | Patients will be enrolled for 18 months and will be followed for 24 months
Event free survival. | Patients will be enrolled for 18 months and will be followed for 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Franck Nicolini, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Result] Nicolini FE, Etienne G, Dubruille V, Roy L, Huguet F, Legros L, Giraudier S, Coiteux V, Guerci-Bresler A, Lenain P, Cony-Makhoul P, Gardembas M, Hermet E, Rousselot P, Ame S, Gagnieu MC, Pivot C, Hayette S, Maguer-Satta V, Etienne M, Dulucq S, Rea D, Mahon FX. Nilotinib and peginterferon alfa-2a for newly diagnosed chronic-phase chronic myeloid leukaemia (NiloPeg): a multicentre, non-randomised, open-label phase 2 study. Lancet Haematol. 2015 Jan;2(1):e37-46. doi: 10.1016/S2352-3026(14)00027-1. Epub 2015 Jan 7. PMID 26687426